CLINICAL TRIAL: NCT04187066
Title: Goal-directed and Cue-dependent Behavior in Severe Obesity
Acronym: PIT_BS
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Sabine Frank, Reserach Associate, University Hospital Tuebingen
Other Study IDs: PIT_BS
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Eating Behavior; Habits; Obesity
MeSH Terms: conditions — Feeding Behavior; Habits; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Obese: severe obesity
  Interventions: Behavioral: mindset induction
- Control: Control group with normal weight
  Interventions: Behavioral: mindset induction

INTERVENTIONS:
Behavioral: mindset induction — induction of a health mindset to measure changes in cue-dependent and goal-directed behavior

SUMMARY:
The current proposal aims to investigate implicit and explicit priming paradigms for changing cue-dependent and goal-directed nutritional behavior in participants with severe obesity before and after bariatric surgery as well as in a control group with normal weight.

DETAILED DESCRIPTION:
Food choice and intake is a daily and throughout normal subject. However, for more and more people eating habits and the question of food choice are of increasing interest and in several cases even a problem. The prevalence of obesity has tripled in the last decades and it is even spoken of an obesity epidemic. Life style interventions to lose weight often fail on the long run, also because people fall back into former unhealthy eating habits. Bariatric surgery is a very effective procedure to reduce weight fundamentally.

Various factors influence our daily food choice, not all of which are apparent to ourselves. Thus, food choice might be goal-directed and therefore conscious and reflective, yet in other circumstances the choice to eat something specific might be based on cue dependent processes which are automatic and thus difficult to control. The aim of the current study is to investigate cue-dependent and goal-directed nutritional behavior as well as the effect of a health mindset induction in severe obesity as well as changes in such behaviors due to bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* experimental: severe obesity
* control: normal weight

Exclusion Criteria:

* impaired cognitive functions, which might conflict with the task
* appropriate German

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * experimental: severe obesity who might get a bariatric surgery
  * control: normal weight
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
changes in food choice behavior due to substantial weight loss by bariatric surgery | pre bariatric surgery, 1 month after bariatric surgery, 6 months after bariatric surgery
  changes in cue-dependent and goal-directed food choices assessed by the Pavlovian-to-instrumental transfer task

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Tuebingen, fMEG Center, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No